CLINICAL TRIAL: NCT00750750
Title: Efficacy and Safety of 200 mcg QD or 200 mcg BID Mometasone Furoate Nasal Spray (MFNS) vs Amoxicillin vs Placebo as Primary Treatment of Subjects With Acute Rhinosinusitis
Brief Title: Effectiveness and Safety of Once or Twice Daily Mometasone Nasal Spray Versus Amoxicillin Versus Placebo for Treatment of Acute Rhinosinusitis (Study P02683)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P02683
Record Dates: First submitted 2008-09-10; First posted 2008-09-11 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Acute Rhinosinusitis
MeSH Terms: interventions — Mometasone Furoate; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- 1 (Active Comparator): MFNS once daily
  Interventions: Drug: mometasone furoate nasal spray (MFNS)
- 2 (Experimental): MFNS twice daily
  Interventions: Drug: MFNS
- 3 (Active Comparator): Amoxicillin
  Interventions: Drug: Amoxicillin
- 4 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: mometasone furoate nasal spray (MFNS) — Placebo capsules three times daily for 10 days, and MFNS 50 mcg/spray, 2 sprays in each nostril once daily in the morning and placebo nasal spray once daily in the evening for 15 days, followed by 14-day no-treatment observation period
  Other Names: SCH 32088; Nasonex
  Arms: 1
Drug: MFNS — Placebo capsules three times daily for 10 days, and MFNS 50 mcg/spray, 2 sprays in each nostril twice daily for 15 days followed by 14-day no-treatment observation period
  Other Names: SCH 32088; Nasonex
  Arms: 2
Drug: Amoxicillin — Amoxicillin 500 mg/capsule, one capsule 3 times a day for 10 days and placebo nasal spray twice daily for 15 days, followed by a 14-day no-treatment observation period
  Arms: 3
Drug: Placebo — Placebo capsule three times daily for 10 days and placebo nasal spray twice daily for 15 days, followed by 14-day no-treatment observation
  Arms: 4

SUMMARY:
This study was conducted to compare the effectiveness and safety of mometasone nasal spray once daily or twice daily with amoxicillin or with placebo in treating the signs and symptoms of acute rhinosinusitis. Patients received mometasone nasal spray 2 sprays per nostril once daily, 2 sprays per nostril twice daily, amoxicillin 500 mg three times a day, or placebo three times a day. Patients on nasal spray were treated for 15 days and patients on amoxicillin or placebo were treated for 10 days. All patients were followed-up with a 14-day no-treatment observation period.

ELIGIBILITY:
Inclusion Criteria:

Subjects must:

* have been diagnosed with acute rhinosinusitis
* have had signs and symptoms of rhinosinusitis for at least 7 but not more than 28 days prior to Baseline
* have had a major symptom score >=5 and <=12 at the Screening and Baseline, and no more than 3 of the 5 major individual symptoms were to be rated as "severe"
* be >=12 years old
* be in good health overall and normal laboratory tests
* not be pregnant, intending to become pregnant or intending to impregnate.

Exclusion Criteria:

Subjects who:

* have a history of chronic rhinosinusitis or who had undergone sinus or nasal surgery for chronic rhinosinusitis in the 6 months prior to Screening
* have fever >=101°F and/or persistent severe unilateral facial pain/tooth pain; and/or orbital or peri-orbital facial swelling; and/or dental involvement; and/or worsening symptoms after initial improvement
* have a history of symptomatic seasonal allergic rhinitis who were exposed to allergenic pollens
* have asthma with FEV1<65% of predicted volume in the past 3 months or who have had an exacerbation within the past 30 days
* have nasal polyps, Kartagener's syndrome, and otitis or atrophic rhinitis
* have certain comorbid conditions or contraindications to certain drug therapies

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 981 (Actual)
Dates: Start 2003-01-01 (Actual); Primary Completion 2003-09-01 (Actual); Study Completion 2003-09-01 (Actual)

PRIMARY OUTCOMES:
Average AM/PM major-symptom score (sum of rhinorrhea, post nasal drip, nasal congestion/stuffiness, sinus headache, and facial pain/pressure/tenderness on palpation over the paranasal sinuses) over the Treatment Phase of 15 days. | Over 15 days

SECONDARY OUTCOMES:
The total-, major-, and individual-symptom scores (for AM, PM, and AM/PM average) by week, and for Days 1-15, and 16-29. | At end of each week, over Days 1-15, and Days 16-29
Time to onset of action in the major-symptom score, defined as the first day active treatment was statistically significantly different from placebo, and sustained thereafter. | Throughout the Treatment Period
Global response between the groups at Visit 4 or the last treatment visit | At Visit 4 or the last treatment visit
Proportion of subjects who were considered by the investigator to be treatment failures, and proportion of subjects who discontinued early due to treatment failure | Throughout the study

REFERENCES:
- [Result] Meltzer EO, Bachert C, Staudinger H. Treating acute rhinosinusitis: comparing efficacy and safety of mometasone furoate nasal spray, amoxicillin, and placebo. J Allergy Clin Immunol. 2005 Dec;116(6):1289-95. doi: 10.1016/j.jaci.2005.08.044. Epub 2005 Oct 24. PMID 16337461